CLINICAL TRIAL: NCT07126639
Title: A Study on the Short-course Treatment Regimen Containing Pretomanid for Drug-resistant Tuberculosis
Acronym: BPaLM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan Pulmonary Hospital (Other)
Responsible Party: Principal Investigator, Yan Hu, Wuhan Pulmonary hospital, Wuhan Pulmonary Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wuhan Pulmonary H
Record Dates: First submitted 2025-07-13; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Efficacy and Safety
Keywords: BPaLM; short-course treatment regiment
MeSH Terms: interventions — bedaquiline; pretomanid; Linezolid; Moxifloxacin; OPC-67683; Fumigant 93; Levofloxacin; Clofazimine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- test group (Experimental): A six - month regimen containing bedaquiline (BDQ), pretomanid (Pa), linezolid (LZD), and moxifloxacin (MFX)
  Interventions: Drug: bedaquiline; Drug: Pretomanid (Pa); Drug: linezolid; Drug: Moxifloxacin (M)
- Control group (Group A) (Active Comparator): The control group was stratified according to the drug susceptibility results of fluoroquinolones (FQs). The FQs - sensitive group was treated with the BDLL regimen (bedaquiline (BDQ), delamanid (DLM), linezolid (LZD), and levofloxacin (LFX)), the FQs - resistant group was treated with the BDLC regimen (BDQ, DLM, LZD, and clofazimine (CFZ)), and the group with unknown drug susceptibility was treated with the BDLLfxC regimen (BDQ, DLM, LZD, LFX, and CFZ). The duration of all regimens was 6 months.
  Interventions: Drug: bedaquiline; Drug: linezolid; Drug: Delamanid (D); Drug: Levofloxacin; Drug: clofazimine

INTERVENTIONS:
Drug: bedaquiline — Administer 400 mg orally once daily for the first two weeks, followed by 200 mg orally three times a week for the subsequent 22 weeks.
Drug: Pretomanid (Pa) — Administer 200 mg orally once daily for six months.
  Arms: test group
Drug: linezolid — Administer 600 mg orally once daily for six months.
Drug: Moxifloxacin (M) — Administer 400 mg orally once daily for six months.
  Arms: test group
Drug: Delamanid (D) — Administer 100 mg orally twice daily for six months.
  Arms: Control group (Group A)
Drug: Levofloxacin — Administer 800 mg orally once daily for six months.
  Arms: Control group (Group A)
Drug: clofazimine — Administer 100 mg orally once daily for six months.
  Arms: Control group (Group A)

SUMMARY:
Rifampicin-resistant tuberculosis (RR-TB) is characterized by a long treatment course, high incidence of adverse reactions, low cure rate and high recurrence rate. This is related to the large number of drugs in the RR-TB treatment regimen, high incidence of adverse reactions and long treatment course, which leads to poor patient compliance. There is an urgent need for new, effective and safe short-course regimens for drug-resistant tuberculosis. A 6-month short-course oral regimen containing pretomanid was introduced in 2020. However, as pretomanid is not yet available in China, it has not been verified and promoted in China. Pretomanid is expected to be launched in China in 2025, and it is urgent to evaluate the application of the new short-course regimen containing pretomanid in the Chinese population. This study is a prospective, randomized, controlled clinical trial. It plans to include RR-TB patients aged ≥12 years in multiple domestic centers. Under the guidance of rapid molecular drug susceptibility test results, the experimental group will be treated with bedaquiline, pretomanid, linezolid and moxifloxacin for 6 months, while the control group will be treated with bedaquiline, delamanid, linezolid and levofloxacin or bedaquiline, delamanid, linezolid and clofazimine for 6 months, depending on the susceptibility to fluoroquinolones. For patients with unknown susceptibility to fluoroquinolones, bedaquiline, delamanid, linezolid, levofloxacin and clofazimine will be used for 6 months. The efficacy and safety will be evaluated to provide a basis for the introduction and implementation of new short-course regimens for RR-TB in China.

DETAILED DESCRIPTION:
Study Design Type This study is a prospective, randomized controlled trial aimed at evaluating the efficacy and safety of different treatment regimens for patients with drug-resistant tuberculosis (RR-TB).

Study Subjects Patients with MDR/RR-TB who meet the inclusion and exclusion criteria will be enrolled in this study. Deviation from the inclusion and exclusion criteria is not allowed as it may compromise the scientific integrity, regulatory acceptability, or safety of the study participants. Therefore, it is crucial to adhere to the criteria specified in the study protocol.

Study Population Study Population: Male or female patients aged ≥12 years, with newly diagnosed or retreated pulmonary tuberculosis, and no contraindications to the study drugs.

Planned Enrollment 200 cases, 100 cases in each group. Inclusion and Exclusion Criteria

Inclusion Criteria:

The study participant (or their legal guardian if the participant lacks legal capacity) voluntarily signs the informed consent form before enrollment.

The study participant (and their guardian) indicates willingness to complete all study steps and intervention cycles.

Male or female, aged ≥12 years, and weighing ≥30 kilograms. Confirmed pulmonary tuberculosis by microbiological diagnosis, with molecular or phenotypic drug susceptibility test results within the last 3 months confirming rifampicin resistance, and confirmed by sputum culture results at enrollment.

For women of childbearing age, not pregnant, willing to undergo a pregnancy test with a negative result, and willing to use highly effective contraceptive measures from signing the informed consent until 3 months after the end of the study treatment.

For men of childbearing age, using condoms or other methods to ensure effective contraception for their sexual partners.

Women who are breastfeeding are willing to stop breastfeeding from signing the informed consent until 3 months after the end of the study treatment.

Willing to undergo HIV testing, and if the result is positive, willing to receive antiretroviral therapy.

Exclusion Criteria:

Previous treatment with bedaquiline (BDQ) or delamanid (DLM) for more than 28 days.

Concurrent hematogenous disseminated pulmonary tuberculosis or severe extrapulmonary tuberculosis (including gastrointestinal tuberculosis, genitourinary tuberculosis, bone and joint tuberculosis, tuberculous meningitis, etc.) as determined by the investigator.

Currently using prohibited drugs as specified in the study protocol, and the investigator believes that the priority of continuing the drug is higher than participating in this study from the perspective of patient benefit.

Known hypersensitivity to any drug in the study protocol. Currently participating in any other drug clinical trial. Cardiovascular disease risk at screening: QTcF interval > 480 milliseconds; history of clinically significant arrhythmia within 60 days before enrollment as determined by the investigator, and the investigator believes that participation in the study may increase the risk; decompensated heart failure; grade 3 hypertension and not reaching the control target; thyroid dysfunction; abnormal serum calcium, magnesium, or potassium levels.

History of optic neuropathy or peripheral neuropathy, and the investigator believes that progression/deterioration may occur during the study or the participant is not suitable for the study.

Liver disease manifestations at screening: active viral hepatitis; decompensated liver cirrhosis.

Kidney disease history or related manifestations at screening: unstable or rapidly progressive kidney disease; moderate/severe renal impairment or end-stage renal disease; male serum creatinine ≥ 133 μmol/L, female serum creatinine ≥ 124 μmol/L.

Other laboratory abnormalities: hemoglobin level < 8.0 g/dL; platelet count < 75,000/mm³; absolute neutrophil count < 1000/mm³; aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 3×ULN; total bilirubin > 2×ULN, or > 1.5×ULN with other liver enzyme abnormalities; albumin < 30 g/L. Researchers believe that study participants are unable to complete the study process or that participation in the study is unsafe for the participants.

Study Process

This study plans to include RR-TB patients aged ≥12 years. Under the guidance of rapid molecular drug susceptibility test results for fluoroquinolones (FQs), patients will be randomly divided into two groups:

Experimental group: treated with a regimen of bedaquiline, pretomanid, linezolid, and moxifloxacin for 6 months.

Control group:

For FQ-sensitive patients, treated with a regimen of bedaquiline, delamanid, linezolid, and levofloxacin for 6 months.

For FQ-resistant patients, treated with a regimen of bedaquiline, delamanid, linezolid, and clofazimine for 6 months.

For patients with unknown FQ susceptibility results, treated with a regimen of bedaquiline, delamanid, linezolid, levofloxacin, and clofazimine for 6 months.

The study duration includes the screening period, treatment period, post-treatment follow-up period, and extended follow-up period. The study treatment is selected based on FQ susceptibility results. Patients with negative sputum culture at 16 weeks continue for 24 weeks, and those with positive sputum culture continue for 36 weeks. Visit frequency: every 4 weeks during the treatment period and every 8 weeks during the post-treatment follow-up period.

Observation Indicators

Outcome and endpoint definitions:

Benign outcomes during the treatment period:

Cure: completing 80% or more of the required medication dose within 28 weeks after the start of study treatment, with no evidence of treatment failure, and negative MTB culture in the last two sputum specimens (collected at least 14 days apart) at the end of treatment.

Completion of treatment: completing 80% or more of the required medication dose within 28 weeks after the start of study treatment, with no evidence of treatment failure, but no evidence of negative MTB culture in two sputum specimens collected at least 14 days apart at the end of treatment.

Benign outcomes during the post-treatment follow-up period:

Cure: negative MTB sputum culture at 72 weeks after enrollment. Negative sputum culture at the last visit before loss to follow-up: if lost to follow-up before 72 weeks after enrollment and the last MTB sputum culture before loss to follow-up is negative.

Benign outcomes during the extended follow-up period:

Cure: negative MTB sputum culture at 108 weeks after enrollment. Negative sputum culture at the last visit before loss to follow-up: if lost to follow-up before 108 weeks after enrollment and the last MTB sputum culture before loss to follow-up is negative.

Adverse outcomes:

Death: death due to any cause. Drug change: permanent replacement or addition of at least one drug due to any reason, except for adjustments based on baseline drug susceptibility.

Drug discontinuation: interruption of at least one drug for more than 14 consecutive days within 16 weeks after the start of study treatment for any reason; after 16 weeks, if sputum culture has turned negative, interruption of drugs is not considered an adverse outcome.

Treatment failure: positive MTB culture in the last two independently collected sputum specimens (collected at least 14 days apart) at the end of treatment.

Extended treatment: continuing anti-tuberculosis treatment after 28 weeks of treatment initiation.

Loss to follow-up: if a study participant fails to attend two consecutive visits within 16 weeks after the start of study treatment, they are considered lost to follow-up; after 16 weeks, if two consecutive visits are missed and sputum culture has not turned negative, they are considered lost to follow-up; if sputum culture has turned negative, it is considered unassessable.

Relapse: if a study participant has a benign outcome at the end of the treatment period but is subsequently diagnosed with RR/MDR/XDR-TB and requires treatment (with evidence that the relapse is caused by RR, MDR, or XDR-TB strains).

Sample size determination Based on the results of the BEAT TB study and current practice, the historical control data for the rate of benign outcomes is set at 75% (the latest success rate for drug-resistant tuberculosis treatment published by the WHO is 63%, but set according to clinical practice in China). The estimated treatment success rate for the treatment group is 86%. Setting a one-sided α = 0.025, Power = 80%, and assuming a dropout rate of 10%, at least 100 participants are needed in each group. Informed Consent Situation

Study participants were screened and recruited by the trial team members at each center during clinical diagnosis and treatment. Those who met the inclusion and exclusion criteria signed the informed consent form with the trial team members at each center. The informed consent form must be approved by experts and the ethics committee from all parties. When signing, the detailed information about the clinical trial must be explained to the study participants, including:

The researcher or their representative will explain the nature of the study to the study participant or their legal authorized representative/guardian, including the purpose of the trial, the process and duration of the trial, examination procedures, the expected benefits and risks for the study participant, inform the study participant that they may be assigned to different groups in the trial, and answer all questions related to the study.

It must be informed to the study participant or their legal authorized representative/guardian that participation in the study is voluntary.

ELIGIBILITY:
Inclusion Criteria:

he research participants themselves voluntarily signed the informed consent form before being enrolled; for those without full capacity for civil conduct, the consent form was signed by their legal guardians.

The research participants (and their guardians) indicated their willingness to complete all steps and intervention periods of the study.

Male or female, aged 12 years or older, weighing 30 kilograms or more. Confirmed cases of pulmonary tuberculosis pathogen, with molecular or phenotypic drug sensitivity results within the past 3 months confirming resistance to rifampicin, and confirmed by the pathogen culture results of sputum collected at the time of enrollment.

Fertile women not in pregnancy, voluntarily undergoing pregnancy tests, with negative results, and willing to use highly effective contraceptive measures from the time of signing the informed consent until 3 months after the end of the study treatment.

For fertile men, use condoms or other methods to ensure effective contraception for their sexual partners.

Women in lactation, willing to stop breastfeeding from the time of signing the informed consent until 3 months after the end of the study treatment.

Voluntary to undergo HIV testing. If the result is positive, voluntarily accept antiretroviral therapy.

Exclusion Criteria:

Had a known hypersensitivity reaction to any drug in the protocol. Was participating in any clinical trial of other drugs. At the screening stage, had cardiovascular disease risk: QTcF interval over 480 milliseconds; within 60 days before enrollment, had a history of clinically significant arrhythmia that the investigator considered could be clinically significant, and the investigator considered that participating in the study might increase the risk; decompensated heart failure; grade 3 hypertension and not reaching the control target; thyroid dysfunction; abnormal serum calcium, magnesium or potassium levels.

Had a history of optic nerve or peripheral nerve lesion, and the investigator considered that it might progress/deteriorate during the study or was not suitable for participating in this study.

At the screening stage, had the following liver disease manifestations: active viral hepatitis; decompensated stage of liver cirrhosis.

At the screening stage, had the following kidney disease history or kidney-related manifestations: unstable or rapidly progressive kidney disease history; moderate/severe renal function impairment or end-stage renal disease; male serum creatinine ≥ 133 μmol/L, female serum creatinine ≥ 124 μmol/L.

Other laboratory test abnormalities: hemoglobin level < 8.0 g/dL; platelet count < 75,000/mm³; absolute neutrophil count < 1000/mm³; aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 3×ULN; total bilirubin > 2×ULN, or > 1.5×ULN, combined with other liver enzyme abnormalities; albumin < 30 g/L.

The investigator considered that the study participants could not complete the study process, or participating in the study was unsafe for the study participants.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Favorable outcomes during the treatment period | From the initiation of treatment until the 28th week.
  Cure: Completing 80% or more of the medication dosage as required by the protocol within 28 weeks after the start of the research treatment, with no evidence of treatment failure, and the Mycobacterium tuberculosis (MTB) cultures of the last two sputum specimens (collection interval ≥ 14 days) at the end of treatment being negative.
  Treatment completion: Completing more than 80% of the medication dosage as required by the protocol within 28 weeks after the start of the research treatment, with no evidence of treatment failure, but without evidence that the MTB cultures of two sputum specimens collected at an interval of at least 14 days are negative.

SECONDARY OUTCOMES:
Favorable outcomes during the follow - up period after treatment | From the beginning of the treatment until 72 weeks.
  Cure: Negative Mycobacterium tuberculosis (MTB) sputum culture at 72 weeks after enrollment.
  Negative sputum culture at the last visit before loss to follow - up: If the patient is lost to follow - up before 72 weeks after enrollment and the last MTB sputum culture before loss to follow - up is negative.
Favorable outcomes with an extended follow - up period | Follow - up was conducted until 108 weeks after enrollment.
  Cure: Negative mycobacterium tuberculosis (MTB) sputum culture at 108 weeks after enrollment.
  Negative sputum culture at the last visit before loss to follow - up: If the patient is lost to follow - up before 108 weeks after enrollment and the last MTB sputum culture before loss to follow - up is negative.
Unfavorable outcome | From the time of enrollment until the 108th week of follow - up
  Death: Occurrence of death due to any cause. Drug replacement: Permanent replacement or addition of at least one medication due to any reason, excluding adjustments based on baseline drug susceptibility.
  Drug discontinuation: Discontinuation of at least one medication for more than 14 consecutive days within 16 weeks after the initiation of the study treatment for any reason; after 16 weeks, if sputum conversion has occurred, drug discontinuation is not considered an adverse outcome.
  Treatment failure: At the end of treatment, the results of Mycobacterium tuberculosis (MTB) culture from the last two independently collected sputum specimens (with a collection interval of ≥14 days) are positive.
  Extended treatment: Continuation of anti - tuberculosis treatment after 28 weeks from the start of treatment.
  Loss to follow - up: A study participant is considered lost to follow - up if they miss two consecutive follow - up visits within 16 weeks after the initiation of the study treatment; af

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Wei, M.D., Study Director — Wuhan Pulmonary Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code